CLINICAL TRIAL: NCT04354701
Title: The COVID-19 and Cancer Consortium (CCC19) Registry
Brief Title: COVID-19 and Cancer Consortium Registry
Acronym: CCC19
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Jeremy Warner, Principal Investigator, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC MD 2032
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: COVID-19; Invasive Malignancy (Any Type)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Web-based REDCap survey — The survey takes approximately 5-10 minutes to complete and includes five parts: 1) basic demographics about the patient, including performance status and comorbidities; 2) initial COVID-19 diagnosis and clinical course; 3) cancer and cancer treatment details; 4) respondent details; 5) long-term COVID-19 outcomes.

SUMMARY:
In this study we will collect granular information on cancer patients infected with COVID-19, as rapidly as possible. The mechanism for collection of this information is a de-identified centralized registry housed at Vanderbilt University Medical Center, with data donations from internal and external health care professionals.

DETAILED DESCRIPTION:
The COVID-19 and Cancer Consortium (CCC19) registry prospectively collects anonymized data about patients diagnosed with COVID-19 and cancer. The goal of the registry is to generate hypothesis-generating and hypothesis-supporting findings that are generalizable to the population at large. Specifically:

I. Characterize patient factors, such as pre-existing comorbidities, baseline medication exposures, cancer type, status, and treatment, and demographic factors that are associated with short- and long-term outcomes of COVID-19 (laboratory-confirmed or presumptive), including severity and fatality, in patients with cancer.

II. Describe cancer treatment modifications made in response to COVID-19, including dose adjustments, changes in symptom management, or temporary or permanent cessation.

III. Evaluate the association of COVID-19 with cancer outcomes.

ELIGIBILITY:
Inclusion criteria:

• Healthcare providers or their proxies who would like to report a patient with ALL of the following criteria:

* Suspected (presumptive positive based on clinical presentation) or lab-confirmed COVID-19.
* Current or past medical history of invasive malignancy (any type)

Exclusion criteria:

* Participants at international sites not explicitly listed below
* Non-healthcare providers (or their proxies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the COVID-19 and Cancer Consortium (CCC19).
Sampling Method: Non-Probability Sample
Enrollment: 19275 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Web-based REDCap survey | Approximately 18 months
  The survey includes five parts: 1) basic demographics about the patient, including performance status and comorbidities; 2) initial COVID-19 diagnosis and clinical course; 3) cancer and cancer treatment details; 4) respondent details; 5) long-term COVID-19 outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Warner, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Nagaraj G, Vinayak S, Khaki AR, Sun T, Kuderer NM, Aboulafia DM, Acoba JD, Awosika J, Bakouny Z, Balmaceda NB, Bao T, Bashir B, Berg S, Bilen MA, Bindal P, Blau S, Bodin BE, Borno HT, Castellano C, Choi H, Deeken J, Desai A, Edwin N, Feldman LE, Flora DB, Friese CR, Galsky MD, Gonzalez CJ, Grivas P, Gupta S, Haynam M, Heilman H, Hershman DL, Hwang C, Jani C, Jhawar SR, Joshi M, Kaklamani V, Klein EJ, Knox N, Koshkin VS, Kulkarni AA, Kwon DH, Labaki C, Lammers PE, Lathrop KI, Lewis MA, Li X, Lopes GL, Lyman GH, Makower DF, Mansoor AH, Markham MJ, Mashru SH, McKay RR, Messing I, Mico V, Nadkarni R, Namburi S, Nguyen RH, Nonato TK, O'Connor TL, Panagiotou OA, Park K, Patel JM, Patel KG, Peppercorn J, Polimera H, Puc M, Rao YJ, Razavi P, Reid SA, Riess JW, Rivera DR, Robson M, Rose SJ, Russ AD, Schapira L, Shah PK, Shanahan MK, Shapiro LC, Smits M, Stover DG, Streckfuss M, Tachiki L, Thompson MA, Tolaney SM, Weissmann LB, Wilson G, Wotman MT, Wulff-Burchfield EM, Mishra S, French B, Warner JL, Lustberg MB, Accordino MK, Shah DP; COVID-19 and Cancer Consortium. Clinical characteristics, racial inequities, and outcomes in patients with breast cancer and COVID-19: A COVID-19 and cancer consortium (CCC19) cohort study. Elife. 2023 Oct 17;12:e82618. doi: 10.7554/eLife.82618. PMID 37846664
- [Derived] Moey MYY, Hennessy C, French B, Warner JL, Tucker MD, Hausrath DJ, Shah DP, DeCara JM, Bakouny Z, Labaki C, Choueiri TK, Dent S, Akhter N, Ismail-Khan R, Tachiki L, Slosky D, Polonsky TS, Awosika JA, Crago A, Wise-Draper T, Balanchivadze N, Hwang C, Fecher LA, Gomez CG, Hayes-Lattin B, Glover MJ, Shah SA, Gopalakrishnan D, Griffiths EA, Kwon DH, Koshkin VS, Mahmood S, Bashir B, Nonato T, Razavi P, McKay RR, Nagaraj G, Oligino E, Puc M, Tregubenko P, Wulff-Burchfield EM, Xie Z, Halfdanarson TR, Farmakiotis D, Klein EJ, Robilotti EV, Riely GJ, Durand JB, Hayek SS, Kondapalli L, Berg S, O'Connor TE, Bilen MA, Castellano C, Accordino MK, Sibel B, Weissmann LB, Jani C, Flora DB, Rudski L, Dutra MS, Nathaniel B, Ruiz-Garcia E, Vilar-Compte D, Gupta S, Morgans A, Nohria A; COVID-19 and Cancer Consortium. COVID-19 severity and cardiovascular outcomes in SARS-CoV-2-infected patients with cancer and cardiovascular disease. Transl Oncol. 2023 Aug;34:101709. doi: 10.1016/j.tranon.2023.101709. Epub 2023 Jun 2. PMID 37302348
- [Derived] Bakouny Z, Labaki C, Grover P, Awosika J, Gulati S, Hsu CY, Alimohamed SI, Bashir B, Berg S, Bilen MA, Bowles D, Castellano C, Desai A, Elkrief A, Eton OE, Fecher LA, Flora D, Galsky MD, Gatti-Mays ME, Gesenhues A, Glover MJ, Gopalakrishnan D, Gupta S, Halfdanarson TR, Hayes-Lattin B, Hendawi M, Hsu E, Hwang C, Jandarov R, Jani C, Johnson DB, Joshi M, Khan H, Khan SA, Knox N, Koshkin VS, Kulkarni AA, Kwon DH, Matar S, McKay RR, Mishra S, Moria FA, Nizam A, Nock NL, Nonato TK, Panasci J, Pomerantz L, Portuguese AJ, Provenzano D, Puc M, Rao YJ, Rhodes TD, Riely GJ, Ripp JJ, Rivera AV, Ruiz-Garcia E, Schmidt AL, Schoenfeld AJ, Schwartz GK, Shah SA, Shaya J, Subbiah S, Tachiki LM, Tucker MD, Valdez-Reyes M, Weissmann LB, Wotman MT, Wulff-Burchfield EM, Xie Z, Yang YJ, Thompson MA, Shah DP, Warner JL, Shyr Y, Choueiri TK, Wise-Draper TM; COVID-19 and Cancer Consortium. Interplay of Immunosuppression and Immunotherapy Among Patients With Cancer and COVID-19. JAMA Oncol. 2023 Jan 1;9(1):128-134. doi: 10.1001/jamaoncol.2022.5357. PMID 36326731
- [Derived] Grivas P, Khaki AR, Wise-Draper TM, French B, Hennessy C, Hsu CY, Shyr Y, Li X, Choueiri TK, Painter CA, Peters S, Rini BI, Thompson MA, Mishra S, Rivera DR, Acoba JD, Abidi MZ, Bakouny Z, Bashir B, Bekaii-Saab T, Berg S, Bernicker EH, Bilen MA, Bindal P, Bishnoi R, Bouganim N, Bowles DW, Cabal A, Caimi PF, Chism DD, Crowell J, Curran C, Desai A, Dixon B, Doroshow DB, Durbin EB, Elkrief A, Farmakiotis D, Fazio A, Fecher LA, Flora DB, Friese CR, Fu J, Gadgeel SM, Galsky MD, Gill DM, Glover MJ, Goyal S, Grover P, Gulati S, Gupta S, Halabi S, Halfdanarson TR, Halmos B, Hausrath DJ, Hawley JE, Hsu E, Huynh-Le M, Hwang C, Jani C, Jayaraj A, Johnson DB, Kasi A, Khan H, Koshkin VS, Kuderer NM, Kwon DH, Lammers PE, Li A, Loaiza-Bonilla A, Low CA, Lustberg MB, Lyman GH, McKay RR, McNair C, Menon H, Mesa RA, Mico V, Mundt D, Nagaraj G, Nakasone ES, Nakayama J, Nizam A, Nock NL, Park C, Patel JM, Patel KG, Peddi P, Pennell NA, Piper-Vallillo AJ, Puc M, Ravindranathan D, Reeves ME, Reuben DY, Rosenstein L, Rosovsky RP, Rubinstein SM, Salazar M, Schmidt AL, Schwartz GK, Shah MR, Shah SA, Shah C, Shaya JA, Singh SRK, Smits M, Stockerl-Goldstein KE, Stover DG, Streckfuss M, Subbiah S, Tachiki L, Tadesse E, Thakkar A, Tucker MD, Verma AK, Vinh DC, Weiss M, Wu JT, Wulff-Burchfield E, Xie Z, Yu PP, Zhang T, Zhou AY, Zhu H, Zubiri L, Shah DP, Warner JL, Lopes G. Association of clinical factors and recent anticancer therapy with COVID-19 severity among patients with cancer: a report from the COVID-19 and Cancer Consortium. Ann Oncol. 2021 Jun;32(6):787-800. doi: 10.1016/j.annonc.2021.02.024. Epub 2021 Mar 19. PMID 33746047
- [Derived] Kuderer NM, Choueiri TK, Shah DP, Shyr Y, Rubinstein SM, Rivera DR, Shete S, Hsu CY, Desai A, de Lima Lopes G Jr, Grivas P, Painter CA, Peters S, Thompson MA, Bakouny Z, Batist G, Bekaii-Saab T, Bilen MA, Bouganim N, Larroya MB, Castellano D, Del Prete SA, Doroshow DB, Egan PC, Elkrief A, Farmakiotis D, Flora D, Galsky MD, Glover MJ, Griffiths EA, Gulati AP, Gupta S, Hafez N, Halfdanarson TR, Hawley JE, Hsu E, Kasi A, Khaki AR, Lemmon CA, Lewis C, Logan B, Masters T, McKay RR, Mesa RA, Morgans AK, Mulcahy MF, Panagiotou OA, Peddi P, Pennell NA, Reynolds K, Rosen LR, Rosovsky R, Salazar M, Schmidt A, Shah SA, Shaya JA, Steinharter J, Stockerl-Goldstein KE, Subbiah S, Vinh DC, Wehbe FH, Weissmann LB, Wu JT, Wulff-Burchfield E, Xie Z, Yeh A, Yu PP, Zhou AY, Zubiri L, Mishra S, Lyman GH, Rini BI, Warner JL; COVID-19 and Cancer Consortium. Clinical impact of COVID-19 on patients with cancer (CCC19): a cohort study. Lancet. 2020 Jun 20;395(10241):1907-1918. doi: 10.1016/S0140-6736(20)31187-9. Epub 2020 May 28. PMID 32473681